CLINICAL TRIAL: NCT05667545
Title: Evaluation of the Remineralizing Effect of Self-assembling Peptide P11-4 on Caries Affected Dentin.
Brief Title: Evaluation of the Effect of Self-Assembling Peptide P11-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nafesa Mostafa
Record Dates: First submitted 2022-12-12; First posted 2022-12-28 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Peptides; P11-4 peptide

STUDY DESIGN:
Intervention Model Description: To study the effect of self assembling-peptide P11-4 treatment on dentine remineralization, after removal of all infected dentine (Remineralization of caries affected dentin),
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative control group (A1) (Active Comparator): A1: cavities will be sealed directly by restorative material (conventional glass ionomer) without any treatment.
  Interventions: Drug: Peptide
- Treatment group (A2) (Active Comparator): A2: cavities will be treated by Self-Assembling peptide P11-4 then sealed by conventional glass ionomer.
  Interventions: Drug: Peptide

INTERVENTIONS:
Drug: Peptide — it is about synthetic protein acting on tooth structure help information apatite crystals
  Other Names: peptide P11-4

SUMMARY:
Dental caries is a biofilm-mediated, sugar-driven, multifactorial, dynamic disease that results in the phasic demineralization and remineralization of dental hard tissues.

These tissues have poor regeneration capability because of the lack of both regenerative cells and vascularization.

In the complex caries progression process involving dietary sugars, bacterial metabolism and demineralization, the collagenous organic matrix becomes exposed and destroyed by resident and bacterial proteases, allowing the lesion to expand

DETAILED DESCRIPTION:
It is possible to find numerous noninvasive or minimally invasive therapies for caries such as hygiene education, fluorides, Phosphopeptide compounds, xylitol and infiltrative resins.

However, when caries progresses to the point of breaking down the dental tissues, composite restorations are imperative to preserve the tooth functionality.

During the execution of routine dental restorations, the hybrid structure formed by the dental bonding procedure occurs through the interaction and subsequent polymerization of monomers around the demineralized collagen matrix.

The oral cavity is a severe environment for the resin-dental bond to survive for a reasonable length of time, with thermomechanical changes, chemical attacks by acids and enzymes and other factors posing routine daily challenges. Therefore to achieve effective and stable bonding, the preservation of dentin collagen is critical, since collagen represents the major organic component of the dentin matrix.

Based on today's understanding of the dental biomineralization process, new efforts have been made to develop synthetic analogues of non-collagenous proteins (NCPs), which are involved in the events of nucleation and growth of hydroxyapatite crystals in hard tissues Such analogues have been designed mirroring the amphiphilic characteristics of NCPs, with polar groups complexing inorganic ions and non-polar side chains governing the matrix-matrix interactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study will be required to present at least one permanent molar with an active deep carious lesion without pulpal involvement.
* Age of patient: 18 -30 years
* Carious lesions will be standardized by means of clinical and radiographic examinations performed before the procedures

Exclusion Criteria:

* Teeth with deep dentinal lesions with pulpal involvement, abscess, pain or swelling
* Developmental disorders and adjacent soft tissue lesions
* Patients with systemic illness will be excluded

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Remineralization | 3 months
  Assessment of the remineralizing effect of self-assembling peptide P11-4 on affected-caries dentin. Remineralization will be assessed by radiodensity using digital radiography

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Mosleh, Lecturer, Principal Investigator — Al-Azhar Faculty of Dentistary for girls
Locations (1):
- Faculty of Dentistary - Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided